CLINICAL TRIAL: NCT06125834
Title: Trastuzumab Emtansine (T-DM1) Treatment in HER2-positive Breast Cancer Patients With Progressive Disease After TKIs or HP Therapy: a Multicenter, Single-arm, Phase II Study
Brief Title: Trastuzumab Emtansine (T-DM1) in HER2-positive Breast Cancer Patients With Progressive Disease After TKIs or HP Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJMU-BC02
Record Dates: First submitted 2023-10-29; First posted 2023-11-09 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Advanced Breast Cancer; Objective Response Rate; Trastuzumab Emtansine
MeSH Terms: interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T-DM1 treatment group (Experimental): Trastuzumab Emtansine (T-DM1), 3.6mg/kg, d1/21, IVD, until progressive diseases or intolerable adverse effects occurs
  Interventions: Drug: Trastuzumab Emtansine (T-DM1)

INTERVENTIONS:
Drug: Trastuzumab Emtansine (T-DM1) — Enrolled patients will receive Trastuzumab Emtansine (T-DM1) treatment (3.6mg/kg, d1/21, IVD) until progressive diseases or intolerable adverse effects occurs.

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of trastuzumab emtansine (T-DM1) in the treatment of patients with advanced HER2-positive breast cancer after TKIs or HP therapy. The main questions it aims to answer are:

* The objective response rate of patients receiving T-DM1 therapy with advanced HER2-positive breast cancer after TKIs or HP therapy.
* The adverse events and prognosis of patients with advanced HER2-positive breast cancer who receive the T-DM1 therapy.
* Changes of anti-tumor immunity during T-DM1 therapy in patients with advanced HER2-positive breast cancer.

Participants will receive T-DM1 treatment (3.6mg/kg, d1/21, IVD) until progressive diseases or intolerable adverse effects occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; pregnancy test (-) for premenopausal and perimenopausal patients, promising to use reliable contraception during treatment.
* Patients who were be diagnosed with invasive breast cancer according to the eighth edition of American Joint Committee on Cancer (AJCC) staging system, and develop disease progression after anti-HER2 therapy (TKIs) for stage IV disease at initial diagnosis or within one year of adjuvant anti-HER2 therapy (HP) after surgery for early breast cancer.
* At least one measurable lesion according to RECIST 1.1.
* ECOG score of 0 or 1.
* The organ function is still good and meets the following indicators: hemoglobin ≥ 90g/L, white blood cell ≥ 3.5×10^9/L, platelet ≥ 100×10^9/L, neutrophil ≥ 1.5×10^9/L, aspartate aminotransferase or alanine aminotransferase ≤ 3×ULN, total bilirubin ≤ 1.5×ULN, serum creatinine value ≤ 1.5×ULN.
* Without myocardial ischemia in ECG.
* NYHA grade I; Echocardiography LVEF ≥55%; Cardiac markers: cardiac troponin (cTnI) and brain natriuretic peptide (BNP) within normal range.
* Complete all necessary baseline laboratory and radiological tests prior to treatment.
* Complete clinical data.

Exclusion Criteria:

* male breast cancer or inflammatory breast cancer.
* Patients who have other malignant tumors or have contracted malignant tumors other than breast cancer in the past 5 years, except for basal cell carcinoma of the skin or flat cell carcinoma and carcinoma in situ of the cervix that have been adequately treated and controlled.
* Accompanying other anti-tumor treatments or participating in other clinical trials.
* Serious diseases that will affect the patient's compliance or put the patient at risk.
* Major surgical procedures performed within 4 weeks prior to the commencement of study treatment or anticipated major surgical procedures during the course of the study.
* Patients who have used ADC drugs at present or before this study.
* History of allergic reactions or contraindications to use of any drug ingredient in this study.
* Patients with chronic diarrhea and intestinal obstruction, as well as other diseases that affect drug administration and absorption.
* Patients who have clinical cardiac symptoms or diseases that are not well controlled, such as: heart failure above NYHA 2; unstable angina; myocardial infarction occurred within one year; clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
* Dementia, intellectual abnormality, or any mental illness that interferes with the understanding of informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 12 months

SECONDARY OUTCOMES:
Progression-free survival | up to 36 months
Overall survival | up to 36 months
Adverse events | every 6 weeks
Antitumor immunity related parameters | up to 12 weeks
  The changes of composition and function of immune cells in the tumor and peripheral blood before and after treatment
Tumor related parameters | up to 12 weeks
  Tumor heterogeneity before and after treatment its correlation with objective response rate, progression-free survival, overall survival, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- JiangSu Province Hospital/ The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Wolff AC, Hammond ME, Hicks DG, Dowsett M, McShane LM, Allison KH, Allred DC, Bartlett JM, Bilous M, Fitzgibbons P, Hanna W, Jenkins RB, Mangu PB, Paik S, Perez EA, Press MF, Spears PA, Vance GH, Viale G, Hayes DF; American Society of Clinical Oncology; College of American Pathologists. Recommendations for human epidermal growth factor receptor 2 testing in breast cancer: American Society of Clinical Oncology/College of American Pathologists clinical practice guideline update. J Clin Oncol. 2013 Nov 1;31(31):3997-4013. doi: 10.1200/JCO.2013.50.9984. Epub 2013 Oct 7. PMID 24101045
- [Background] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012
- [Background] Swain SM, Miles D, Kim SB, Im YH, Im SA, Semiglazov V, Ciruelos E, Schneeweiss A, Loi S, Monturus E, Clark E, Knott A, Restuccia E, Benyunes MC, Cortes J; CLEOPATRA study group. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA): end-of-study results from a double-blind, randomised, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Apr;21(4):519-530. doi: 10.1016/S1470-2045(19)30863-0. Epub 2020 Mar 12. PMID 32171426
- [Background] Peddi PF, Hurvitz SA. Trastuzumab emtansine: the first targeted chemotherapy for treatment of breast cancer. Future Oncol. 2013 Mar;9(3):319-26. doi: 10.2217/fon.13.7. PMID 23469968
- [Background] Hunter FW, Barker HR, Lipert B, Rothe F, Gebhart G, Piccart-Gebhart MJ, Sotiriou C, Jamieson SMF. Mechanisms of resistance to trastuzumab emtansine (T-DM1) in HER2-positive breast cancer. Br J Cancer. 2020 Mar;122(5):603-612. doi: 10.1038/s41416-019-0635-y. Epub 2019 Dec 16. PMID 31839676
- [Background] Verma S, Miles D, Gianni L, Krop IE, Welslau M, Baselga J, Pegram M, Oh DY, Dieras V, Guardino E, Fang L, Lu MW, Olsen S, Blackwell K; EMILIA Study Group. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med. 2012 Nov 8;367(19):1783-91. doi: 10.1056/NEJMoa1209124. Epub 2012 Oct 1. PMID 23020162
- [Background] Krop IE, Kim SB, Gonzalez-Martin A, LoRusso PM, Ferrero JM, Smitt M, Yu R, Leung AC, Wildiers H; TH3RESA study collaborators. Trastuzumab emtansine versus treatment of physician's choice for pretreated HER2-positive advanced breast cancer (TH3RESA): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):689-99. doi: 10.1016/S1470-2045(14)70178-0. Epub 2014 May 2. PMID 24793816
- [Background] Ding S, Chen X, Shen K. Single-cell RNA sequencing in breast cancer: Understanding tumor heterogeneity and paving roads to individualized therapy. Cancer Commun (Lond). 2020 Aug;40(8):329-344. doi: 10.1002/cac2.12078. Epub 2020 Jul 12. PMID 32654419
- [Background] Gao Y, Wu N, Wang S, Yang X, Wang X, Xu B. Concurrent mutations associated with trastuzumab-resistance revealed by single cell sequencing. Breast Cancer Res Treat. 2021 Jun;187(3):613-624. doi: 10.1007/s10549-021-06237-0. Epub 2021 Apr 27. PMID 33905021